CLINICAL TRIAL: NCT02132195
Title: Adrenocorticotropic Hormone (ACTH) for Frequently Relapsing and Steroid Dependent Nephrotic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Larry Greenbaum, MD, PhD, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00068101; EmoryPedNeph-002 (Other: Emory Division of Pediatric Nephrology)
Record Dates: First submitted 2013-12-12; First posted 2014-05-07 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Adrenocorticotropic hormone (ACTH) (Active Comparator): Patients will receive ACTH twice weekly subcutaneously The initial dosing will be based on body surface area (BSA): 80 IU/1.73 m2
  The patients will receive the initial dose for 6 months. At 6 months, the dose will be reduced by 50%. Patients who have side effects may have the dose reduced by 50% during the initial 6 months. A second dose reduction would still occur at 6 months (25% of initial dose).
  Interventions: Drug: ACTH
- No treatment (No Intervention): Patients in this treatment arm will receive no treatment to prevent relapses of nephrotic syndrome. A relapse, if it occurs, will be treated with prednisone and the patient will leave the no treatment arm of the study.
- Rescue therapy (Active Comparator): There is an option for the patient in no-treatment arm to elect to be placed in the active treatment arm of the trial (rescue therapy).
  Interventions: Drug: ACTH

INTERVENTIONS:
Drug: ACTH — Patients will receive ACTH twice weekly for 6 months, with a 50% dose reduction allowed for side effects. The dose will be reduce by 50% at 6 months and continued for an additional 6 months.
  Other Names: Acthar; Adrenocorticotropic hormone
  Arms: Adrenocorticotropic hormone (ACTH); Rescue therapy

SUMMARY:
In childhood nephrotic syndrome, the kidneys leak protein, causing body swelling and a variety of possible complications such as infection, blood clots, and kidney failure. The first-line treatment for nephrotic syndrome is corticosteroids. Many children respond to prednisone treatment, but the disease comes back (relapses) when the prednisone is stopped or the dose is reduced. Children with frequently relapsing or steroid dependent nephrotic syndrome are at risk for toxicity from frequent exposure to corticosteroids.

Currently, the standard treatment for frequently relapsing and steroid dependent nephrotic syndrome involves a variety of medications that suppress the immune system, which can produce serious side effects. We propose a study to examine the effects of a different medication, ACTH, on nephrotic syndrome. ACTH is a hormone naturally found in the body. Recently, in adult studies, ACTH has been shown to be effective for the treatment of nephrotic syndrome. It has also been shown to have mild and reversible side effects. ACTH is potentially an attractive therapeutic alternative for the treatment of frequently relapsing and steroid dependent nephrotic syndrome in children. Our study will randomly assign patients with frequently relapsing or steroid dependent nephrotic syndrome to either ACTH treatment or no treatment. This will allow us to study the effects of ACTH on this disease and its side effects, by comparing how patients do on ACTH treatment versus no treatment. We hypothesize that ACTH gel is superior to no treatment in maintaining remission in children with frequently relapsing or steroid dependent nephrotic syndrome.

DETAILED DESCRIPTION:
Our hypotheses are the following:

Hypothesis 1: ACTH gel is superior to no treatment in maintaining remission in children with frequently relapsing or steroid dependent nephrotic syndrome (NS).

Hypothesis 2: Relapses in children with frequently relapsing or steroid dependent nephrotic syndrome receiving ACTH gel will increase when the dose of ACTH gel is reduced by 50%.

Hypothesis 3: ACTH gel will increase the percentage of children with frequently relapsing or steroid dependent nephrotic syndrome that remain relapse free off medication.

Primary end-points:

The primary end-point related to Hypothesis 1 is the proportion of patients in each arm with a relapse during the initial 6 months of treatment.

The primary end-point related to Hypothesis 2 is the proportion of relapse-free patients during the first 6 months and second 6 months of treatment with ACTH. This will include patients initially randomized to ACTH and patients who receive ACTH as rescue therapy following their initial relapse in patients randomized to no treatment.

The primary end-point related to Hypothesis 3 is the proportion of patients who have relapses in the 6 months following completion of one year of ACTH. This will be compared to the proportion of patients with relapses during the initial 6 months in the patients randomized to no treatment.

Secondary end-points:

Our secondary end-points are the following:

1. The total prednisone exposure over the initial 12 months in the two groups.
2. The number of relapses over the initial 6 months in the two groups.
3. The change in body mass index (BMI), height standard deviation score (SDS), and cholesterol over the study period for both groups Study Design and Methods The experimental design is a multi-center, prospective, controlled open label, randomized trial comparing ACTH gel and no treatment in preventing relapses in pediatric patients with frequently relapsing or steroid dependent nephrotic syndrome.

Patients will be randomized in a 1:1 ratio to either no treatment or treatment with ACTH gel. The primary outcome will be the presence of a relapse within 6 months of starting ACTH gel or no treatment.

After initial recruitment, enrollment will begin with a screening visit to determine eligibility and obtain informed consent and assent. Randomization and weaning of all other medications for the treatment of NS will begin after remission has been achieved for those with active relapse. There will be a 2 week overlap of ACTH and current immunosuppressive medications:

1. ACTH will be initiated 2 weeks prior to the completion of the prednisone taper for patients who are receiving prednisone at the time of consent.
2. ACTH will be initiated 2 weeks prior to stopping preventive medications such as tacrolimus, cyclosporin, and mycophenolate.

Patients randomized to no treatment will be followed for up to 6 months or until disease relapse, whichever occurs first. Patients who relapse within 6 months will be given the option of reassignment to the ACTH treatment group after remission has been achieved using conventional corticosteroid therapy.

Patients randomized to ACTH treatment will be given ACTH for 12 months. During the second 6 months, the ACTH dose will be reduced to 50% of the starting dose. The outcome of interest is the presence of relapses after dose reduction. Follow-up will occur throughout the 12 months of therapy, and also for 6 months following the completion of ACTH therapy. The outcome of interest is the percentage of patients with relapses in the 6 months after completing a 12 month course of ACTH treatment.

The primary end-point of the study and on which the statistical power is based is the proportion of patients who have a relapse in the 6 months following randomization to either ACTH or no ACTH.

We hypothesize that the 6 month relapse rate for patients receiving no treatment is 70%. In order to detect a 6 month relapse rate of 30% for patients receiving the ACTH gel, we will randomize 30 patients in each arm using a two sided z test with alpha=.05. Our statistical power to detect such a difference is 91% which assumes two interim analyses at 50% and 100% of accumulated information. That is, once 30 patients have 6 month relapse data, we will conduct the first interim analysis. The last one will be completed once we have relapse data on all 60 patients. The table below gives the operating characteristics for such a design:

Number of Patients with 6 Months Data Boundary p-value 30 0.006 60 0.045

Using the method of Lan-DeMets, we list the boundary p-value for this sequential design. Thus, after our first interim look, we will reject the null hypothesis of equal 6 month relapse rates between ACTH gel and no treatment if our test statistic renders a p-value < .006. According to the intent to treat principle, patients will be analyzed according to the treatment they have been assigned to during the randomization procedure. The odds ratio of ACTH versus no ACTH, plus the Wald 95% confidence interval, will be also be calculated.

The primary end-point related to specific aim 2 is the proportion of relapse-free patients during the first 6 months and second 6 months of treatment with ACTH. This will include patients initially randomized to ACTH and patients who receive ACTH as rescue therapy following their initial relapse. We will estimate 6 month and 12 month relapse-free rate using the method of Kaplan-Meier and compare treatments using a log-rank test.

The primary end-point related to specific aim 3 is the proportion of patients who have relapses in the 6 months following completion of one year of ACTH. This will be compared to the proportion of patients with relapses during the initial 6 months in the patients randomized to no treatment using a z test statistic. Odds ratios of ACTH vs no ACTH will also be calculated.

We will also compare patients as randomized by secondary endpoints such as total prednisone exposure in 12 months, number of relapses, cholesterol and change in BMI with two sample t-tests. If normality assumptions do not hold, appropriate non-parametric methods will be used.

Growth data collected during the study will be summarized descriptively for each treatment group at each time point. Based on height data collected during the study and published reference height information, the height standard deviation score (SDS, also called z-score) will be computed for each patient at each time point as:

(Height - mean height for that age category) / SD of height for that age category.

Descriptive statistics of this endpoint will be presented by time point and the z-scores will allow identification of potential outliers.

Treatment Assignment and Randomization Treatment assignments will be stratified according to clinical center. The treatment assignments will be generated by the Data Coordinating Center (DCC) with the use of a pseudo-random-number generator with randomly permutated blocks that will be used to ensure balance between the number of subjects assigned to each treatment (ACTH or no ACTH). Before the study starts, the institutional research coordinator at each clinical center will be given a batch of 20 sealed, sequenced, opaque envelopes containing the treatment assignment and will have a unique identification number consisting of the clinical center stratum.

Patients will be assigned to one of the two treatment arms in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Age >1 year at onset of nephrotic syndrome
2. Age 2-20 years at time of randomization
3. Estimated glomerular filtration rate (GFR) > 50 ml/min/1.73 m2 at most recent measure prior to randomization (Schwartz formula)
4. Steroid responsive nephrotic syndrome throughout clinical course (never required a second agent to attain remission of a relapse of nephrotic syndrome)
5. History of frequently relapsing or steroid dependent nephrotic syndrome (defined as 2 or more relapses within 6 months after initial therapy or 4 or more relapses in any 12 month period OR relapse during taper or within 2 weeks of discontinuing prednisone).
6. Patient is currently in relapse of nephrotic syndrome or had a relapse within the last 4 months (defined as an increase in the first morning urine protein to creatinine ratio ≥2 or Albustix reading of ≥2 for 3 or 5 consecutive days).

Exclusion Criteria:

1. Prior treatment with ACTH.
2. Cyclophosphamide or rituximab within the last 4 months.
3. Lactation, pregnancy, or refusal of birth control in females with child-bearing potential
4. Planned treatment with live or live-attenuated vaccines once enrolled in the study.
5. Participation in another therapeutic trial concurrently or 30 days prior to randomization
6. Active/serious infection (including, but not limited to Hepatitis B or C, HIV)
7. Malignancy concurrently or within the last 2 years.
8. Blood pressure >95% for age/height while receiving maximal doses of 3 or more medications.
9. Prior diagnosis of diabetes mellitus (Type I or II) or fasting glucose >200mg/dL
10. Organ transplantation
11. Contraindications to Acthar: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenal cortical hyperfunction
12. Secondary cause of nephrotic syndrome (e.g., SLE)
13. Biopsy demonstrating a diagnosis other than minimal change, focal segmental glomerulosclerosis (FSGS) or a variant (mesangial proliferation, Immunoglobulin M nephropathy)
14. Inability to consent/assent -

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Greenbaum, MD, PhD, Principal Investigator — Emory University
Locations (16):
- United States (16):
  - Pediatric Nephrology of Alabama, PC., Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - Nemours/AI duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Boston Children's Hopsital, Boston, Massachusetts
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy, Kansas City, Missouri
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke Children's Health Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of Richmond at VCU, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 31 patients enrolled: 15 were randomized to receive ACTH, and 16 were randomized to No-treatment. There was an option for patients in No-treatment arm to elect to be placed on ACTH (rescue therapy). 13 patients in No-treatment arm used this option, and received ACTH as rescue therapy.
Groups:
- Adrenocorticotropic Hormone (ACTH): Patients will receive ACTH twice weekly subcutaneously The initial dosing will be based on body surface area (BSA): 80 IU/1.73 m2
  The patients will receive the initial dose for 6 months. At 6 months, the dose will be reduced by 50%. Patients who have side effects may have the dose reduced by 50% during the initial 6 months. A second dose reduction would still occur at 6 months (25% of initial dose).
  ACTH: Patients will receive ACTH twice weekly for 6 months, with a 50% dose reduction allowed for side effects. The dose will be reduce by 50% at 6 months and continued for an additional 6 months.
- No Treatment: Patients in this treatment arm will receive no treatment to prevent relapses of nephrotic syndrome. A relapse, if it occurs, will be treated with prednisone and the patient will leave the no treatment arm of the study. There is an option for the patient to elect to be placed in the active treatment arm of the trial (rescue therapy).
- Rescue Therapy: Patients moved from No-treatment group to receive rescue ACTH therapy twice weekly for 6 months, with a 50% dose reduction allowed for side effects. The dose will be reduce by 50% at 6 months and continued for an additional 6 months.
  Other Names: Acthar Adrenocorticotropic hormone
Period: Initial Assignment
Arm/Group | Adrenocorticotropic Hormone (ACTH) | No Treatment | Rescue Therapy
Started | 15 | 16 | 0
Completed | 1 | 16 | 0
Not Completed | 14 | 0 | 0
Not completed — Relapsed | 14 | 0 | 0
Period: Rescue Therapy
Arm/Group | Adrenocorticotropic Hormone (ACTH) | No Treatment | Rescue Therapy
Started (There was an option for No-treatment pts to be placed on ACTH (rescue therapy). 13 pts used it) | 0 | 0 | 13
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 11
Not completed — Relapsed | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adrenocorticotropic Hormone (ACTH) | No Treatment | Rescue Therapy | Total
Number analyzed (Participants) | 15 | 16 | 13 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Of 31 patients enrolled: 15 were randomized to receive ACTH, and 16 were randomized to No-treatment. There was an option for patients in No-treatment arm to elect to be placed on ACTH (rescue therapy). 13 patients in No-treatment arm used this option, and received ACTH as rescue therapy.
  years
    Initial assignment: number analyzed (Participants) | 15 | 16 | 0 | 31
    Initial assignment | 7.0 [4.8 to 11.2] | 9.5 [5.2 to 12.0] |  | 8.6 [4.3 to 12.9]
    Rescue therapy: number analyzed (Participants) | 0 | 0 | 13 | 13
    Rescue therapy |  |  | 9.15 [4.84 to 11.9] | 9.15 [4.84 to 11.9]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Of 31 patients enrolled: 15 were randomized to receive ACTH, and 16 were randomized to No-treatment. There was an option for patients in No-treatment arm to elect to be placed on ACTH (rescue therapy). 13 patients in No-treatment arm used this option, and received ACTH as rescue therapy.
  Participants
    Initial assignment: number analyzed (Participants) | 15 | 16 | 0 | 31
    Initial assignment: Female | 5 | 4 | 0 | 9
    Initial assignment: Male | 10 | 12 | 0 | 22
    Rescue therapy: number analyzed (Participants) | 0 | 0 | 13 | 13
    Rescue therapy: Female |  |  | 3 | 3
    Rescue therapy: Male |  |  | 10 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Of 31 patients enrolled: 15 were randomized to receive ACTH, and 16 were randomized to No-treatment. There was an option for patients in No-treatment arm to elect to be placed on ACTH (rescue therapy). 13 patients in No-treatment arm used this option, and received ACTH as rescue therapy.
  Participants
    Initial assignment: number analyzed (Participants) | 15 | 16 | 0 | 31
    Initial assignment: American Indian or Alaska Native | 0 | 0 |  | 0
    Initial assignment: Asian | 0 | 1 |  | 1
    Initial assignment: Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Initial assignment: Black or African American | 2 | 1 |  | 3
    Initial assignment: White | 13 | 13 |  | 26
    Initial assignment: More than one race | 0 | 0 |  | 0
    Initial assignment: Unknown or Not Reported | 0 | 1 |  | 1
    Rescue therapy: number analyzed (Participants) | 0 | 0 | 13 | 13
    Rescue therapy: American Indian or Alaska Native |  |  | 0 | 0
    Rescue therapy: Asian |  |  | 1 | 1
    Rescue therapy: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
    Rescue therapy: Black or African American |  |  | 0 | 0
    Rescue therapy: White |  |  | 12 | 12
    Rescue therapy: More than one race |  |  | 0 | 0
    Rescue therapy: Unknown or Not Reported |  |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Initial assignment | 15 | 16 | 0 | 31
  United States: Rescue therapy | 0 | 0 | 13 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experienced a Relapse of Nephrotic Syndrome
Description: Number of participants experienced a relapse of nephrotic syndrome during the initial 6 months of the study.
Time Frame: 6 months
Population: The primary outcome measure was accessed during the initial 6 months based on initial assignment, rescue therapy group was not part of the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Rescue Therapy: Patients moved from No-treatment group to receive rescue ACTH therapy twice weekly for 6 months, with a 50% dose reduction allowed for side effects. The dose will be reduce by 50% at 6 months and continued for an additional 6 months.
  Other Names:
  Acthar Adrenocorticotropic hormon
Arm/Group | Adrenocorticotropic Hormone (ACTH) | No Treatment | Rescue Therapy
Number analyzed (Participants) | 15 | 16 | 0
Participants | 14 | 15 |

2. Secondary Outcome: Number of Participants Experiencing Relapses After Dose Reduction of ACTH
Description: The dose of ACTH will be reduced by 50% after 6 months and the rate of relapse during this period will be evaluated.
Time Frame: 6 to 12 months
Population: Three participants who completed 6 months of ACTH Full Dose therapy and then 6 months of Reduced Dose ACTH - inclusive of one subject initially randomized to ACTH and two subjects who received ACTH as rescue treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Adrenocorticotropic Hormone (ACTH) | No Treatment | Rescue Therapy
Number analyzed (Participants) | 1 | 0 | 2
Participants | 0 |  | 0

3. Secondary Outcome: Number of Adverse Events
Description: Adverse events will be collected (SAEs and AEs)
Time Frame: 12 months
Population: 15 pts randomized to receive ACTH, and 16 pts randomized to No-treatment. 13 patients in No-treatment arm elected to receive ACTH as rescue therapy.
Measure: Number; unit: number of events
Arm/Group | Adrenocorticotropic Hormone (ACTH) | No Treatment | Rescue Therapy
Number analyzed (Participants) | 15 | 16 | 13
number of events | 12 | 4 | 17

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Adrenocorticotropic Hormone (ACTH) | No Treatment | Rescue Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/16 | 2/13
Other Adverse Events (participants affected / at risk) | 4/15 | 2/16 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adrenocorticotropic Hormone (ACTH) (N=15) | No Treatment (N=16) | Rescue Therapy (N=13)
Hospitalization for renal disease relapse affecting multiple systems (General disorders) | 3 (5) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adrenocorticotropic Hormone (ACTH) (N=15) | No Treatment (N=16) | Rescue Therapy (N=13)
Flu and strep infections (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Behavioral changes (Social circumstances) | 2 (2) | 0 (0) | 1 (1)
Sleep disturbances (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Increase in blood pressure (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Increase in Cushingoid symptoms (Endocrine disorders) | 0 (0) | 1 (1) | 3 (4)
Swelling, redness, rash at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (5)
Rash under arms (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT02132195/Prot_SAP_000.pdf